CLINICAL TRIAL: NCT01401699
Title: Optical Coherence Tomography Based Screening and Surveillance of Esophagus and Gastroesophageal Junction
Brief Title: Optical Coherence Tomography (OCT) Based Screening of Esophagus and Gastroesophageal Junction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2006-P-000203; 5R21CA141884 (NIH)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's; esophagus; OCT; imaging
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Frequency Domain imaging System (Experimental): Optical Frequency Domain Imaging (OFDI) balloon based imaging
  Interventions: Device: Optical Frequency Domain Imaging (OFDI)

INTERVENTIONS:
Device: Optical Frequency Domain Imaging (OFDI) — Optical Frequency Domain (OFDI) imaging of esophagus

SUMMARY:
The specific aim of this study is to determine the accuracy of Optical Coherence Tomography (OCT) imaging for screening and diagnosis of the distal esophagus in patients undergoing a clinical esophagogastroduodenoscopy (EGD) procedure. The accuracy of results obtained using the developed OCT imaging probe will be determined and compared with those obtained through the traditional standard of care endoscopic biopsy .

DETAILED DESCRIPTION:
Three hundred consenting patients undergoing routine esophagogastroduodenoscopy (EGD) procedures will be recruited for examination at the gastroesophageal junction with our developed OCT imaging system. The patients will undergo a clinical EGD procedure including endoscopic biopsy. The first step in the procedure follows the standard care with the performance of the surveillance endoscopy. The study experimental procedure will then begin. This study requires the use of a balloon . The balloon placement method is in accordance with current standard clinical practice and involves the insertion of a guide wire through the auxiliary channel of the endoscope. The endoscope is then removed, leaving the guide wire in place, and the OCT balloon is inserted the required distance (determined during the endoscopy) over the guide wire to the GE junction. The OCT balloon will then be inflated and will remain in this fixed position throughout the entire procedure. Once the OCT imaging probe is in place, OCT image data will be continuously collected over the length of the balloon(approximately 5 cm).

It is expected that the total examination time including insertion and inflation of the OCT balloon, OCT imaging and removal of the OCT balloon will add no more than 10 minutes to the total length of the EGD.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18,
* capable of giving informed consent,
* are undergoing elective EGD, and
* if female are willing to take a pregnancy test

Exclusion Criteria:

* patients on oral anticoagulation medications,
* with a history of hemostasis disorders and
* patients that are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-09; Primary Completion 2011-11-16 (Actual); Study Completion 2011-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachussetts General Hospital; Norman Nishioka, MD, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Massachussetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Optical Frequency Domain Imaging System: OFDI imaging
  Optical Frequency Domain Imaging (OFDI) System: OFDI Imaging of esophagus
Period: Overall Study
Arm/Group | Optical Frequency Domain Imaging System
Started | 109
Completed | 109
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects completed the study. Imaging was not performed for one subject because of the system malfunction.
Arm/Group | Optical Frequency Domain Imaging System
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Which the Entire Distal Esophagus Can be Visualized Using the Balloon Based Optical Coherence Tomography Screening
Description: Collected entire distal esophagus OFDI Images analyzed and compared to the images obtained during standard of care surveillance endoscopy.
Time Frame: Images will be acquired during the OFDI imaging session which should take an average of 5 minutes
Population: All subjects completed the study with no adverse events.
Measure: Count of Participants; unit: Participants
Groups:
- Optical Frequency Domain Imaging: Optical Frequency Domain imaging data
Arm/Group | Optical Frequency Domain Imaging
Number analyzed (Participants) | 109
Participants | 109

ADVERSE EVENTS:
Time Frame: During the imaging session
Arm/Group | Optical Frequency Domain Imaging System
All-Cause Mortality (participants affected / at risk) | 0/109
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 0/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optical Frequency Domain Imaging System (N=109)
aspiration (Investigations) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No